CLINICAL TRIAL: NCT02401087
Title: The Anaesthesiological Approach to Varicocele Correction in Outpatients Setting: an Observational Analysis
Status: Completed | Type: Observational
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Andrea Luigi Ambrosoli, M.D., Ospedale di Circolo - Fondazione Macchi
Other Study IDs: Var-001
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Varicocele
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Anaesthesiological procedure

SUMMARY:
The aim of this observational study was to evaluate, based on the intraoperative anesthetic that is routinely carried out at the Department of Day Surgery, the difference in timing of the patient's discharge from the hospital (ie when the patient has autonomous demabulation and urination spontaneous) in patients undergoing correction of varicocele according Marmar.

ELIGIBILITY:
Inclusion Criteria:

* Male
* ASA I-II
* No mental alteration

Exclusion Criteria:

* Chronic pain
* Allergies to local anaesthetics, acetaminophen,oppioids
* ASA III - IV
* Postoperative discharge to ICU
* Epatic or renal failure
* Mental status alteration
* Coagulopathy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be identified as potentially were to be enrolled in the preoperative anesthetic visit.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
discharge time | one day
  check the elapsed time between the induction of anesthesia and obtaining discharge criteria, urination and deambulation, from the Department of Day Surgery.

SECONDARY OUTCOMES:
Difference in the onset of acute post-operative pain | four days
Check the occurence of any side effects | three months
Clinical evaluation of patients at 1 and 3 months after surgery (possibility of chronic pain) | three months

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Turconi, MD, Principal Investigator — University Hospital Varese
Locations (1):
- Department of Day Surgery Ospedale di Circolo Varese, Varese, VA, Italy